CLINICAL TRIAL: NCT00146107
Title: Weight Loss and Exercise in Frail Obese Elderly Subjects
Brief Title: Weight Loss and Exercise in Obese, Physically Limited, Older Women and Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Dennis T. Villareal, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AG025501-01 (NIH); R01AG025501 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: obesity; aging; exercise; diet; weight loss; physical function; Obesity in the Elderly
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention)
- 2 (Experimental): Weight loss
  Interventions: Behavioral: Diet
- 3 (Experimental): Exercise
  Interventions: Other: Exercise
- 4 (Experimental): Weight loss and exercise
  Interventions: Other: Weight Loss and Exercise

INTERVENTIONS:
Behavioral: Diet — 10 percent weight loss through diet and behavioral modification
  Arms: 2
Other: Exercise — Multicomponent (resistance, aerobic, balance) exercise three times a week
  Arms: 3
Other: Weight Loss and Exercise — 10% weight loss through diet and exercise plus multicomponent exercise training three times a week
  Arms: 4

SUMMARY:
The purpose of this study is to determine the effect of weight loss and exercise on physical function, body fat and muscle mass, bone strength, and quality of life.

DETAILED DESCRIPTION:
Obesity causes serious medical complications and impairs quality of life. Moreover, in elderly persons, obesity can lead to frailty by exacerbating the decline in strength, endurance, balance and mobility associated with aging and physical inactivity. The primary objectives of the proposed research are to evaluate the independent and combined effects of weight loss and exercise on physical function, body composition, bone and muscle metabolism, and quality of life in frail, obese elderly men and women. The central hypothesis is that in frail obese elderly subjects, weight loss will improve physical function and quality of life, while the addition of exercise will not only augment improvement in these outcomes, but also attenuate the adverse effects of weight loss on bone and muscle masses. To test this hypothesis, 110 elderly (65-85 years old) obese men and women (body mass index [BMI] > 30 kg/m2) with physical frailty will be randomized to 4 treatment groups: 1) control, 2) 10% weight loss, 3) exercise training, and 4) 10% weight loss plus exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI 30 or greater)
* Elderly (age 65 years or older)
* Frailty

Exclusion Criteria:

* Major chronic disease or any condition that would interfere with exercise or dietary restriction, in which exercise or dietary restriction are contraindicated, or that would interfere with interpretation of results.
* Examples include cardiopulmonary disease, unstable disease, severe orthopedic or neuromuscular impairments, dementia, history of malignancy during the past 5 years, or current use of bone acting drugs.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 107 (Actual)
Dates: Start 2005-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
physical function | one year

SECONDARY OUTCOMES:
body composition | one year
muscle protein synthesis | one year
quality of life | one year
cognition and mood | one year
metabolism | one year
bone mineral density | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Villareal DT, Banks M, Siener C, Sinacore DR, Klein S. Physical frailty and body composition in obese elderly men and women. Obes Res. 2004 Jun;12(6):913-20. doi: 10.1038/oby.2004.111. PMID 15229329
- [Derived] Colleluori G, Chen R, Napoli N, Aguirre LE, Qualls C, Villareal DT, Armamento-Villareal R. Fat Mass Follows a U-Shaped Distribution Based on Estradiol Levels in Postmenopausal Women. Front Endocrinol (Lausanne). 2018 Jul 2;9:315. doi: 10.3389/fendo.2018.00315. eCollection 2018. PMID 30013511
- [Derived] Colleluori G, Napoli N, Phadnis U, Armamento-Villareal R, Villareal DT. Effect of Weight Loss, Exercise, or Both on Undercarboxylated Osteocalcin and Insulin Secretion in Frail, Obese Older Adults. Oxid Med Cell Longev. 2017;2017:4807046. doi: 10.1155/2017/4807046. Epub 2017 Aug 23. PMID 28951766
- [Derived] Napoli N, Shah K, Waters DL, Sinacore DR, Qualls C, Villareal DT. Effect of weight loss, exercise, or both on cognition and quality of life in obese older adults. Am J Clin Nutr. 2014 Jul;100(1):189-98. doi: 10.3945/ajcn.113.082883. Epub 2014 Apr 30. PMID 24787497
- [Derived] Shah K, Armamento-Villareal R, Parimi N, Chode S, Sinacore DR, Hilton TN, Napoli N, Qualls C, Villareal DT. Exercise training in obese older adults prevents increase in bone turnover and attenuates decrease in hip bone mineral density induced by weight loss despite decline in bone-active hormones. J Bone Miner Res. 2011 Dec;26(12):2851-9. doi: 10.1002/jbmr.475. PMID 21786319
- [Derived] Villareal DT, Chode S, Parimi N, Sinacore DR, Hilton T, Armamento-Villareal R, Napoli N, Qualls C, Shah K. Weight loss, exercise, or both and physical function in obese older adults. N Engl J Med. 2011 Mar 31;364(13):1218-29. doi: 10.1056/NEJMoa1008234. PMID 21449785